CLINICAL TRIAL: NCT04560868
Title: Development of a mHealth Intervention for Ambivalent Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 1401452; R21CA234003 (NIH)
Record Dates: First submitted 2020-06-15; First posted 2020-09-23 (Actual); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Tobacco Use Disorder; Smoking Cessation; Motivation; Behavior, Smoking
Keywords: mHealth; smoking; smoking cessation; motivation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Device: Control mHealth program; Drug: Nicotine patch
- Experimental (Experimental)
  Interventions: Device: Experimental mHealth program; Drug: Nicotine patch

INTERVENTIONS:
Device: Control mHealth program — The intervention includes a mHealth intervention that is grounded in best practice recommendations for treatment of nicotine dependence.
  Arms: Control
Device: Experimental mHealth program — The intervention includes a mHealth intervention that is grounded in best practice recommendations for treatment of nicotine dependence. Experimental participants also receive additional content designed to motivate smoking reduction/quitting and provide skills training.
  Arms: Experimental
Drug: Nicotine patch — Participants in both arms can earn the ability to request a 2-week supply of over-the-counter nicotine patches. Patches are earned through accumulated use of the assigned mHealth program.

SUMMARY:
The current pilot study will assess the feasibility and acceptability of a novel mHealth app designed for people who are ambivalent about quitting smoking. Results will be used to refine the intervention and plan for a future randomized effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Can speak/read English;
* Current smoker;
* Own and regularly use an eligible smartphone;
* No vision impairments;
* Willing to install and use the study program;
* Willing to use birth control if elect to use nicotine replacement during the study (females);
* Meet definition for ambivalence
* Not actively using treatment

Exclusion Criteria:

* Smoke less than 10 cigarettes per day
* Self-report a lifetime history of dementia, manic depression, bipolar disorder, or schizophrenia;
* Have medical contraindications for nicotine replacement therapy;
* Another household member is enrolled in the study
* Unable to verify contact information
* Fail to install app

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McClure, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.

REFERENCES:
- [Derived] McClure JB, Heffner JL, Krakauer C, Mun S, Klasnja P, Catz SL. Feasibility, Acceptability, and Potential Impact of a Novel mHealth App for Smokers Ambivalent About Quitting: Randomized Pilot Study. JMIR Mhealth Uhealth. 2023 Jun 28;11:e46155. doi: 10.2196/46155. PMID 37379059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began 12/16/2020 and study activities completed 9/27/21. Participants were recruited through two sources: (1) social media ads inviting individuals to email contact study staff to learn more and be screened for eligibility and (2) outreach to people our research waitlist.
Period: Overall Study
Arm/Group | Control | Experimental
Started | 29 | 28
Completed 1-month Self-report Survey | 28 | 21
Completed 3-month Self-report Survey | 26 | 21
Completed App Utilization Period | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 27 | 56
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (9.1) | 47.9 (11.5) | 47.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 28 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 24 | 23 | 47
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes/day] | 17.8 (6.6) | 18.5 (8.7) | 18.2 (7.6)
At least one quit attempt lasting a day or longer in the past 12 months [Count of Participants; unit: Participants] | 7 | 7 | 14
7-day point prevalence abstinence [Count of Participants; unit: Participants] — Positive if the participant abstained from smoking (even a puff) in the past 7 days.
  Participants | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Program Engagement
Description: Number of unique app user-sessions
Time Frame: Assessed at 3-month follow-up
Population: All individuals who installed the app (n = 57).
Measure: Mean (Standard Deviation); unit: User sessions
Arm/Group | Control | Experimental
Number analyzed (Participants) | 29 | 28
User sessions | 7.3 (6.6) | 19.9 (16.2)
Statistical Analysis 1: Comparison: Control vs Experimental; Based on a priori power calculations we had 80% power to detect an average increase of 3.8 log ins in the experimental relative to the control arm; Test type: Equivalence — The point null hypothesis was a difference in expected number of log ins of exactly 0; p < 0.01, Regression, Linear; Mean Difference (Final Values) = 12.73, 95% CI 2-sided [6.41 to 19.05] — mean difference=experimental-control

2. Primary Outcome: Quit Attempt Lasting at Least 24 Hours
Description: At least one intentional smoking quit attempt lasting at least 24 hours. Missing outcomes imputed as not making a quit attempt.
Time Frame: Assessed at 3-month follow-up
Population: All individuals who installed the app (n = 57).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 29 | 28
Participants | 11 | 11
Statistical Analysis 1: Comparison: Control vs Experimental; Based on a priori power calculations, we had 80% power to detect a 33% - 35% increase in the proportion of experimental participants who successfully quit smoking for at least 24 hours relative to controls; Test type: Equivalence — The null hypothesis was a point null of relative risk equal to exactly 1; p = 0.98, Regression, Poisson; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.55 to 1.85] — relative risk=experimental/control

3. Primary Outcome: Not Smoking (Even a Puff) in the Last 7 Days
Description: 7-day point prevalent abstinence: self-report of not smoking, even a puff, in the last 7 days. Missing values were imputed as smoking.
Time Frame: Assessed at 3-month follow-up
Population: All individuals who installed the app (n = 57).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 29 | 28
Participants | 2 | 4
Statistical Analysis 1: Comparison: Control vs Experimental; Based on a priori power calculations, we had 80% power to detect a 28% - 33% increase in 7-day smoking abstinence in the experimental arm relative to the control arm at 3 months; Test type: Equivalence — The null hypothesis was a point null of exactly 0 risk difference between arms; p = 0.35, Regression, Linear; Risk Difference (RD) = 0.08, 95% CI 2-sided [-0.08 to 0.24] — Risk difference = experimental - control

4. Secondary Outcome: Satisfaction With Assigned App
Description: Satisfaction with the overall "content and advice" of the assigned app, rated on a Likert scale from 1="not at all satisfied" to 5="extremely satisfied".
Time Frame: Assessed at 1 month
Population: Responses were assessed among participants who earned at least one utilization badge by the one-month survey. This ensured participants had sufficient interaction with the app to rate their satisfaction with it.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 25 | 19
score on a scale | 3.6 (1.2) | 3.8 (1.0)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The null hypothesis was a point null of exactly 0 difference in expected score between arms; p = 0.40, Regression, Linear; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.35 to 0.87] — mean difference=experimental-control

5. Secondary Outcome: Satisfaction With Assigned App
Description: Satisfaction with the overall "content and advice" of the assigned app on a Likert scale from 1="not at all satisfied" to 5="extremely satisfied".
Time Frame: Assessed at 3 months
Population: Responses were assessed among participants who earned at least one utilization badge by the three-month survey. This was done to ensure participants had sufficient interaction with the app to rate their satisfaction with it.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 23 | 20
score on a scale | 4.0 (1.1) | 4.0 (1.1)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The null hypothesis was a point null of exactly 0 difference in expected score between arms; p = 0.90, Regression, Linear; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.68 to 0.60] — mean difference=experimental-control

6. Secondary Outcome: Helpfulness of Assigned App
Description: Global helpfulness rating calculated as the average helpfulness rating of 8 app features, each rated on a Likert scale from 1="not at all helpful" to 5="extremely helpful".
Time Frame: Assessed at 1 month.
Population: Participants who installed the app, self-reported use of all rated features, rated each feature on follow-up survey, and were confirmed via automated data to have used the app features.
Measure: Mean (Standard Deviation); unit: average scores on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 5
average scores on a scale | 3.2 (1.2) | 3.8 (0.8)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The tested hypothesis was a point null of 0 difference in expected average helpfulness score between arms; p = 0.39, Regression, Linear; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.5 to 1.4] — mean difference=experimental-control

7. Secondary Outcome: Helpfulness of Assigned App
Description: Average helpfulness rating of 8 separate app features, with each feature rated on a Likert scale from 1="not at all helpful" to 5="extremely helpful".
Time Frame: Assessed at 3 months
Population: Individuals who installed the app, responded to questions about helpfulness of each rated feature, self-reported use of each app feature, and based on automated data had sufficient use of the app features to rate their helpfulness at follow-up.
Measure: Mean (Standard Deviation); unit: average scores on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 5 | 5
average scores on a scale | 3.1 (0.6) | 3.6 (0.7)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The tested hypothesis was for a point null of 0 difference in expected average helpfulness score between arms; p = 0.11, Regression, Linear; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.1 to 1.3] — mean difference=experimental-control

8. Secondary Outcome: Program Engagement - Earned Badges
Description: Number of accumulated badge rewards earned from using the assigned app.
Time Frame: Assessed at 1-month follow-up
Population: All individuals who installed the app (n = 57).
Measure: Mean (Standard Deviation); unit: badges
Arm/Group | Control | Experimental
Number analyzed (Participants) | 29 | 28
badges | 5.7 (3.7) | 8.6 (5.8)

9. Secondary Outcome: Program Engagement - Earned Badges
Description: Number of accumulated badge rewards earned from using the assigned app.
Time Frame: Assessed at 3-month follow-up
Population: Includes all individuals who installed the app. Everyone used the app at least once.
Measure: Mean (Standard Deviation); unit: Badges
Arm/Group | Control | Experimental
Number analyzed (Participants) | 29 | 28
Badges | 6.1 (3.5) | 10.1 (6.0)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The null hypothesis was a point null of exactly 0 difference in expected number of badges earned in each arm by 3 months post-baseline; p < 0.01, Regression, Linear; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [1.72 to 6.65] — mean difference=experimental-control

10. Secondary Outcome: Self-efficacy to Quit Smoking
Description: Self-reported confidence in quitting smoking on Likert scale from 1="not at all" to 10="extremely".
Time Frame: Assessed at 1 month
Population: Respondents to the assessed question, which was only asked to those still smoking at follow-up and had installed the app.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 27 | 20
score on a scale | 7.5 (2.3) | 7.4 (2.4)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The null hypothesis was a point null of exactly 0 difference in expected score between arms; p = 0.96, Regression, Linear; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-1.02 to 1.18] — mean difference=experimental-control

11. Secondary Outcome: Self-efficacy to Quit Smoking
Description: Self-reported confidence in quitting smoking on a Likert scale from 1="not at all" to 10="extremely".
Time Frame: Assessed at 3 months
Population: Respondents to the assessed question, which was only asked among individuals who were still smoking at follow-up and had installed the app.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 23 | 17
score on a scale | 7.9 (2.1) | 6.8 (2.7)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The null hypothesis was a point null hypothesis of exactly 0 difference in expected score between the arms; p = 0.31, Regression, Linear; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.55 to 0.66] — mean difference=experimental-control

12. Secondary Outcome: Self-efficacy to Stay Quit
Description: Self-reported confidence in ability to stay quit on a Likert scale from 1="not at all" to 10="extremely".
Time Frame: Assessed at 1 month
Population: Respondents to a question only asked among participants who installed the app and reported they had not smoked in the past 7 days.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 0 | 1
score on a scale |  | 6 (NA) — The Overall Number of Participants Analyzed is 1, so the Standard Deviation was not calculated.

13. Secondary Outcome: Self-efficacy to Stay Quit
Description: Self-reported confidence in ability to stay quit (if no smoking in the past 7 days) on a Likert scale from 1="not at all" to 10="extremely".
Time Frame: Assessed at 3 months
Population: Respondents to question asked among individuals who installed the app and reported not smoking in the past 7 days at 3 month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 1 | 2
score on a scale | 10 (NA) — The Overall Number of Participants Analyzed is 1, so the Standard Deviation was not calculated. | 9 (1.4)

14. Secondary Outcome: Earned and Requested Free Nicotine Replacement Therapy
Description: Earned and requested free nicotine replacement therapy (NRT); free NRT could be earned by earning 6 app utilization badges.
Time Frame: Assessed at 1-month follow-up
Population: All individuals who installed the app (n = 57).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 29 | 28
Participants | 2 | 4

15. Secondary Outcome: Earned and Requested Free Nicotine Replacement Therapy
Description: as for outcome 14
Time Frame: Assessed at 3-month follow-up
Population: Individuals who installed the app (n = 57). Note that free NRT is earned when 6 utilization badges have been earned.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 29 | 28
Participants | 2 | 8
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The point null hypothesis was of the exact same proportion of control and experimental subjects requesting NRT; p = 0.06, Regression, Poisson; Risk Ratio (RR) = 3.9, 95% CI 2-sided [0.9 to 16.9] — RR=experimental/control

16. Secondary Outcome: Quit Attempt Lasting at Least 24 Hours
Description: At least one intentional smoking quit attempt lasting at least 24 hours; non-respondents were assumed to not have a successful quit attempt.
Time Frame: Assessed at 1 month follow-up
Population: Individuals who installed the app (n = 57).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 29 | 28
Participants | 6 | 6
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The null hypothesis was a point null of exactly 0 difference in probability of the outcome between arms; p = 0.99, Regression, Poisson; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.38 to 2.65] — risk ratio=experimental/control

17. Secondary Outcome: Change in Cigarettes/Day
Description: Change in number of cigarettes smoked per day from baseline, calculated as (1 month)-baseline.
Time Frame: Assessed at baseline and 1 month
Population: Individuals who installed the app, returned the 1-month survey, and either responded to this item or reported not smoking in the past 7 days. If they reported not smoking for the past 7 days, number of cigarettes were day were coded as 0.
Measure: Mean (Standard Deviation); unit: Cigarettes/day
Arm/Group | Control | Experimental
Number analyzed (Participants) | 27 | 21
Cigarettes/day
  Baseline 30-day average cigarettes/day | 17.9 (6.8) | 17.6 (8.2)
  Change from baseline in number of cigarettes/day at 1 month (using one-month 7-day average) | -5.1 (5.2) | -3.6 (4.6)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The null hypothesis was a point null of exactly 0 difference in expected change from baseline in number of cigarettes smoked per day between arms; p = 0.30, Regression, Linear; Mean Difference (Net) = 1.39, 95% CI 2-sided [-1.21 to 3.99] — treatment difference=experimental-control, where the outcome for each individual is (one month)-baseline

18. Secondary Outcome: Change in Cigarettes/Day
Description: Change in number of cigarettes smoked per day from baseline, calculated as (3 months)-baseline.
Time Frame: Assessed at baseline and 3 months
Population: Individuals who installed the app, returned the 3-month survey, and either responded to this item or reported not smoking in the past 7 days. If they reported not smoking for the past 7 days, number of cigarettes were day were coded as 0.
Measure: Mean (Standard Deviation); unit: Cigarettes/day
Arm/Group | Control | Experimental
Number analyzed (Participants) | 25 | 21
Cigarettes/day
  Baseline 30-day average cigarettes/day | 17.6 (6.9) | 17.9 (8.0)
  Change in daily average cigarettes/day between baseline and three-month (using 7-day average) | -6.7 (7.9) | -5.2 (7.0)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The null hypothesis was a point null of exactly 0 difference in expected change in daily cigarette usage between arms; p = 0.47, Regression, Linear; Mean Difference (Net) = 1.5, 95% CI 2-sided [-2.51 to 5.5] — treatment effect=experimental-control, where the outcome for each individual is (three month)-baseline

19. Secondary Outcome: Refrain From Smoking (Even a Puff) in the Last 7 Days
Description: 7-day point prevalent abstinence: a self-report of not smoking, even a puff, in the past 7 days. Missing outcomes were imputed as smoking.
Time Frame: Assessed at 1-month follow-up
Population: Individuals who installed the app (n = 57).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 29 | 28
Participants | 0 | 1
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Equivalence — The null hypothesis was risk difference of exactly 0; p = 0.30, Regression, Linear; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.03 to 0.11] — risk difference=experimental-control

ADVERSE EVENTS:
Time Frame: For each participant, adverse events (AE's) were collected over a 3 month period, starting at baseline and ending at 3-month follow-up. Events were monitored continually during this period.
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

LIMITATIONS AND CAVEATS:
The purpose of this pilot was to inform feasibility and acceptability of the experimental app among smokers who were ambivalent about quitting. Data were analyzed among participants who installed the app (n = 57). This pilot study was not powered to provide definitive answers about the efficacy of the intervention in promoting smoking abstinence. A larger trial is needed for this.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT04560868/Prot_SAP_000.pdf